CLINICAL TRIAL: NCT05145413
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Efficacy of Adjunctive KarXT in Subjects With Inadequately Controlled Symptoms of Schizophrenia
Brief Title: A Study to Assess Efficacy and Safety of Adjunctive KarXT in Subjects With Inadequately Controlled Symptoms of Schizophrenia
Acronym: ARISE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Karuna Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CN012-0008; CN012-0008 (Other: Bristol-Myers Squibb Protocol ID); KAR-012 (Other: Karuna Pharmaceuticals Protocol ID)
Record Dates: First submitted 2021-11-23; First posted 2021-12-06 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — xanomeline; trospium chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Drug: KarXT (Experimental)
  Interventions: Drug: Xanomeline and Trospium Chloride Capsules
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Xanomeline and Trospium Chloride Capsules — KarXT 50 mg/20 mg BID KarXT 75mg/20 mg BID KarXT 100mg/20 mg BID KarXT 125mg/30 mg BID
  Arms: Drug: KarXT
Drug: Placebo — Placebo Capsules
  Arms: Placebo

SUMMARY:
This is a Phase 3, 6-week, randomized, double-blind, placebo-controlled, multicenter, outpatient study in subjects with schizophrenia with an inadequate response to their current atypical antipsychotic treatment. The primary objective of the study is to assess the efficacy of adjunctive KarXT (a fixed dose combination of xanomeline and trospium chloride twice daily [BID]) versus placebo in the treatment of subjects with inadequately controlled symptoms of schizophrenia as measured by the Positive and Negative Syndrome Scale (PANSS) Total Score.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is aged ≥18 to <65 years at the time of randomization
2. Subject is capable of providing signed Informed Consent Form before any study assessments will be performed
3. Subject has a primary diagnosis of schizophrenia established by a comprehensive psychiatric evaluation based on the DSM-5 criteria and confirmed by Mini International Neuropsychiatric Interview for Schizophrenia and Psychotic Disorder Studies (MINI) version 7.0.2
4. Subject is currently being treated with stable dosing of monotherapy risperidone, paliperidone, aripiprazole, or their LAIs ziprasidone, lurasidone, or cariprazine and has been taking this treatment with the same dosing regimen for at least 8 weeks at the time of Day 1 (Visit 3)
5. The subject has had at least 1 previous inadequate response to above antipsychotics that was dosed appropriately (within the label) for at least 6 weeks
6. The subject has not required psychiatric hospitalization, incarceration in prison, acute crisis intervention, or other increase in the level of care due to symptom exacerbation within 8 weeks of Screening and is psychiatrically stable in the opinion of the Investigator
7. To be eligible for randomization, subjects need to have detectable levels of background antipsychotic medication (measured at Visit 1)
8. Positive and Negative Syndrome Scale (PANSS) total score ≥ 70 at Screening and randomization
9. Clinical Global Impression-Severity (CGI-S) scale with a score ≥ 4 (moderate) at Screening and randomization
10. PANSS Marder Positive symptom factor ≥ 4 on 2 (or more) items (PANSS items, delusions, hallucinations, grandiosity, suspiciousness and persecution, stereotyped thinking, somatic concern, unusual thought content or lack of judgment and insight), at Screening and randomization
11. Subjects with ≤ 20-point decrease in PANSS Total score between Visit 1 and Visit 3
12. Subject is willing and able to visit the clinic in an outpatient setting for the study duration, follow instructions, and comply with the protocol requirements
13. Body Mass Index (BMI) must be within 18 to 40 kg/m2 (inclusive of both values)
14. Subject resides in a stable living situation in the opinion of the Investigator
15. Subject has identified a reliable informant/ caregiver willing and able to assist with study activities as needed throughout the subject's participation in the study. The informant needs to be physically present at the Baseline visit, but can complete the remaining study visits assessments via phone (as needed and as per local regulations). In Bulgaria, the informant needs to physically present at the Baseline visit and should be physically present at all study visits where the Investigator determines that his/her input would be beneficial.
16. Women of childbearing potential (WOCP), or men whose sexual partners are WOCP, must be able and willing to use at least 1 highly effective method of contraception during the study and for at least 1 menstrual cycle (e.g., 30 days) after the last dose of study drug. Sperm donation is not allowed for 30 days after the final dose of the study drug. A female subject is considered to be a WOCP after menarche and until she is in a postmenopausal state for 12 months or otherwise permanently sterile (for which acceptable methods include hysterectomy, bilateral salpingectomy, or bilateral oophorectomy)

Exclusion Criteria:

1. Any primary DSM-5 disorder other than schizophrenia within 12 months before screening (confirmed using MINI version 7.0.2 at screening)
2. The subject has a history of moderate to severe substance use disorder (other than nicotine) within the past 12 months

   1. A Screening subject with mild substance use disorder within the 12 months before Screening must be discussed with the Medical Monitor before being allowed into the study
   2. Subjects who test positive for cannabis at Screening may be permitted to enroll in consultation with the Medical Monitor if the subject's pattern of use is not indicative of a moderate to severe substance use disorder
3. Subject has a history of treatment-resistant schizophrenia defined as:

   a. Failure to minimally respond to 2 adequate courses of antipsychotic drug (APD) pharmacotherapy Note: Failure to minimally respond is defined as persistence symptoms of moderate severity in 2 or more psychotic symptom domains or persistence of severe symptoms in 1 or more psychotic symptom domains despite adequate dose and duration (6 weeks or longer) of APD treatment.
4. History of symptom instability

   a. > 3 psychiatric hospitalizations over the last 12 months or 2 over the last 6 months
5. Current APD is other than aripiprazole, risperidone, paliperidone, or their LAI versions, ziprasidone, lurasidone, or cariprazine
6. Subjects who are diagnosed with schizophreniform disorder or are experiencing their first treated episode of schizophrenia
7. Significant or severe medical conditions including pulmonary, cardiovascular, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or oncologic disease or any other condition that, in the opinion of the Investigator, could jeopardize the safety of the subject or the validity of the study results

   1. eGFR < 60 mL/min
   2. Alanine transaminase or aspartate transaminase (AST) > 1.5 x upper limit of normal (ULN)
   3. Total bilirubin > 1.5 x ULN (Subjects with Gilbert's syndrome can be included as long as direct bilirubin is ≤ 1.5 x ULN)
8. Subjects with human immunodeficiency virus (HIV), cirrhosis, biliary duct abnormalities, hepatobiliary carcinoma, and/or active hepatic viral infections as indicated by medical history, serologies or LFT results
9. History or high risk of urinary retention, gastric retention, or narrow-angle glaucoma as evaluated by the Investigator
10. History of irritable bowel syndrome (with or without constipation) or any serious constipation requiring treatment within the last 6 months
11. Risk for suicidal behavior during the study as determined by the Investigator's clinical assessment and/or C-SSRS as confirmed by the following:

    1. Answers "Yes" on items 4 or 5 (C-SSRS - ideation) with the most recent episode occurring within the 2 months before Screening or,
    2. Answers "Yes" to any of the 5 items (C-SSRS behavior) with an episode occurring within the 12 months before Screening
12. Clinically significant abnormal finding on the physical examination, medical history, ECG, or clinical laboratory results at Screening
13. Urine toxicology screen is positive for phencyclidine, amphetamines, opiates, cocaine, or alcohol (clinically significant alcohol use in the opinion of the Investigator)
14. Subject is currently taking, or plans to take while in the study, any prohibited concomitant medication.
15. Pregnant, lactating, or less than 3 months postpartum
16. If, in the opinion of the Investigator and/or Sponsor/Medical Monitor subject is unsuitable for enrollment in the study or subject has any finding that, in the view of the Investigator and/or Sponsor/Medical Monitor, may compromise the safety of the subject or affect his/her ability to adhere to the protocol visit schedule or fulfill visit requirements
17. Positive test for coronavirus (COVID-19) within 2 weeks or at Screening
18. Subjects with extreme concerns relating to global pandemics, such as COVID-19, that would obscure ratings or be expected to disrupt adherence to trial procedures
19. Unable to taper and discontinue a concomitant medication that would preclude participation in the double-blind adjunctive treatment (e.g., cannot stop anticholinergic)
20. Subjects with prior exposure to KarXT
21. Subjects who experienced any adverse effects due to xanomeline or trospium
22. Subjects who received investigational product as part of a clinical trial within 3 months of Screening
23. Risk of violent or destructive behavior as per Investigator's judgment that would interfere with subject's participation
24. Current involuntary hospitalization or incarcerationor on parole/probation
25. For all male subjects only, any one of the following:

    1. History of bladder stones
    2. History of recurrent urinary tract infections
    3. Serum prostate specific antigen (PSA) >10 ng/mL
    4. An International Prostate Symptom Score (IPSS) of 5 (almost always) on either item 1, 3, 5, or 6
    5. A sum of scores on IPSS items 1, 3, 5, and 6 of ≥9 Note: IPSS will be required only for male subjects ≥ 45 years of age. Subjects already enrolled in the study will have these assessments at their next clinic visit planned after re-consenting to determine current eligibility.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Actual)
Dates: Start 2021-11-12 (Actual); Primary Completion 2025-03-19 (Actual); Study Completion 2025-03-19 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score at Week 6 | Week 6
  The PANSS is a medical scale used for measuring symptom severity of participants with schizophrenia. The PANSS rating form contains 7 positive symptom scales, 7 negative system scales, and 16 general psychopathology symptom scales. Participants are rated from 1 to 7 on each symptom scale. The total score is the sum of all scales with a minimum score of 30 and a maximum score of 210. A decrease in PANSS total score correlates with an improvement in schizophrenia symptoms.

SECONDARY OUTCOMES:
Change from Baseline in Personal Social Performance (PSP) at Week 6 | Week 6
  The PSP scale assesses functioning using a structured clinical interview across four dimensions: socially useful activities, personal and social relationships, self-care, and disturbing and aggressive behaviors. The PSP provides a score between 1 and 100 using a 6-point severity scale
Change from Baseline in Clinical Global Impression-Severity (CGI-S) at Week 6 | Week 6
  The CGI-S modified asked the clinician 1 question: "Considering your total clinical experience, how mentally ill is the participant at this time?" The clinician's answer rated on the following 7-point scale: 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; 7 = among the most extremely ill participants.
Change from Baseline in Positive and Negative Syndrome Scale (PANSS) Marder Positive symptom factor score at Week 6 | Week 6
  The Positive Marder Factor score is derived from the PANSS and consists of the sum of 4 positive symptom items (P), one negative symptom item (N) and 3 general symptom items (G) (P1. Delusions; P3. Hallucinations; P5. Grandiosity; P6. Suspiciousness and persecution; N7. Stereotyped thinking; G1. Somatic concern; G9. Unusual thought content; G12. Lack of judgment and insight).
Change from Baseline in Positive and Negative Syndrome Scale (PANSS) Marder Negative symptom factor score at Week 6 | Week 6
  The Negative Marder Factor score is derived from the PANSS and consists of the sum of 5 negative symptom items (N) and 2 general symptom items (G) (N1. Blunted affect; N2. Emotional withdrawal; N3. Poor rapport; N4. Passive/apathetic social withdrawal; N6. Lack of spontaneity; G7. Motor retardation; and G16. Active social avoidance), with a minimum score of 7 and a maximum score of 49.
Categorical response defined as the proportion of subjects achieving a ≥ 30% improvement in PANSS total score at Week 6 | Week 6
Preference of Medication (POM) at Week 6 | Week 6
  The POM is a two-item questionnaire assessing the patient's and informant's preference, respectively, for the current antipsychotic as compared with the most recent pre-study antipsychotic. The POM is scored on the following scale: 1 = 'much better, I prefer this medication,' 2 = 'slightly better,' 3 = 'about the same,' 4 = 'slightly worse,' and 5 = 'much worse, I much prefer my previous medication.'

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (166):
- United States (79):
  - IMA Clinical Research, Phoenix, Arizona
  - Local Institution - 147, Phoenix, Arizona
  - Pillar Clinical Research, LLC, Little Rock, Arkansas
  - Woodland International Research Group, LLC, Little Rock, Arkansas
  - Advanced Research Center, Inc., Anaheim, California
  - CITrials - Bellflower, Bellflower, California
  - Synexus Clinical Research US, Inc., Cerritos, California
  - Clinical Innovations Inc., Costa Mesa, California
  - Proscience Research Group, Culver City, California
  - CenExel Collaborative Neuroscience Research, Garden Grove, California
  - Omega Clinical Trials, La Habra, California
  - Sunwise Clinical Research, LLC., Lafayette, California
  - Synergy Clinical Research of Escondido, Lemon Grove, California
  - Encino Hospital Medical Center, Los Angeles, California
  - Excell Research, Inc., Oceanside, California
  - Neuropsychiatric Research Center of Orange County, Orange, California
  - CNRI - Los Angeles, LLC, Pico Rivera, California
  - CenExel Clinical Innovations, Inc., Riverside, California
  - Cnri-San Diego, San Diego, California
  - Stanford University School of Medicine, Stanford, California
  - CenExel Collaborative Neuroscience Research, Torrance, California
  - Local Institution - 186, Coral Gables, Florida
  - Reliable Clinical Research LLC, Hialeah, Florida
  - Galiz Research, LLC, Hialeah, Florida
  - Adaptive Clinical Research, Inc, Lauderhill, Florida
  - Behavioral Clinical Research , Inc, Miami, Florida
  - Premier Clinical Research Institute, Inc., Miami, Florida
  - San Marcus Research Clinic, Inc., Miami Lakes, Florida
  - Assertive Research Center, Miami Lakes, Florida
  - Envision Trials LLC, Miami Springs, Florida
  - Local Institution - 124, Orange City, Florida
  - Pines Care Research Center, Inc., Pembroke Pines, Florida
  - Interventional Psychiatry of Tampa Bay, Tampa, Florida
  - Grady Memorial Hospital, Atlanta, Georgia
  - Synexus Clinical Research US, Inc., Atlanta, Georgia
  - Local Institution - 192, Atlanta, Georgia
  - Local Institution - 135, Augusta, Georgia
  - CenExel iResearch Atlanta, Decatur, Georgia
  - Psych Atlanta, P.C., Marietta, Georgia
  - CenExel iResearch, LLC, Savannah, Georgia
  - Northwestern University, Chicago, Illinois
  - American Medical Research, Inc., Chicago, Illinois
  - Uptown Research Institute, LLC, Chicago, Illinois
  - Phoenix Medical Research, Inc., Prairie Village, Kansas
  - IMA Clinical Research, Monroe, Louisiana
  - CenExel Center for Behavioral Health, Gaithersburg, Maryland
  - Local Institution - 158, Boston, Massachusetts
  - Local Institution - 187, Boston, Massachusetts
  - Local Institution - 185, Worcester, Massachusetts
  - Michigan Clinical Research Institute PC, Ann Arbor, Michigan
  - Cherry Health, Grand Rapids, Michigan
  - Western Michigan University Homer Stryker M.D. School of Medicine, Kalamazoo, Michigan
  - Local Institution - 129, St Louis, Missouri
  - Arch Clinical Trials LLC, St Louis, Missouri
  - Omaha Insomnia and Psychiatric Services LLC, Omaha, Nebraska
  - Altea Research Institute, Las Vegas, Las Vegas, Nevada
  - CenExel Hassman Research Institute, Berlin, New Jersey
  - Synexus Clinical Research US, Inc., New York, New York
  - Manhattan Psychiatric Center, New York, New York
  - Manhattan Behavioral Medicine, PLLC, New York, New York
  - Psychiatry and Alzheimer's Care of Rochester. PLLC, Rochester, New York
  - Richmond Behavioral Associates ERG Clinical Research - New York PLLC, Staten Island, New York
  - Clinical Trials of America - Psychiatry, Hickory, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Local Institution - 168, Garfield Heights, Ohio
  - Insight Clinical Trials LLC, Independence, Ohio
  - The Rivus Wellness & Research Institute, Oklahoma City, Oklahoma
  - Prevention Science Institute, Eugene, Oregon
  - Community Clinical Research, Inc., Austin, Texas
  - InSite Clinical Research; LLC, DeSoto, Texas
  - JPS Health Network, Fort Worth, Texas
  - Ben Taub Hospital, Houston, Texas
  - Clinical Trial Network LLC, Houston, Texas
  - University Hills Clinical Research - Irving, Irving, Texas
  - Pillar Clinical Research, LLC, Richardson, Texas
  - At Health Texas, Richmond, Texas
  - Perceptive Pharma Research, Richmond, Texas
  - Green Mountain Research Institute, Rutland, Vermont
  - Northwest Clinical Research Center, Bellevue, Washington
- Bulgaria (21):
  - MHAT Dr. Hristo Stambolski, EOOD, Kazanlak, Stara Zagora
  - Ambulatory for Individual Practice for Specialized Medical Care in Psychiatry - Dr Ivo Natsov, Cherven Bryag
  - Medical Centre 'Asklepii', OOD, Dupnitsa
  - Medical Center Lifemed, Kardzhali
  - State Psychiatric Hospital 'Sv. Ivan Rilski', Novi Iskar, Novi Iskar
  - Medical Center Medconsult Pleven OOD, Pleven
  - UMHAT 'Dr. Georgi Stranski', EAD, Pleven
  - UMHAT Sv. Georgi, EAD, Plovdiv
  - Local Institution - 321, Plovdiv
  - Local Institution - 313, Razgrad
  - MHAT Dr Ivan Seliminski AD, Sliven
  - Medical Center 'Sv.Naum', Sofia
  - MHC - Sofia, EOOD, Sofia
  - Local Institution - 320, Sofia
  - DCC 'Sv. Vrach and Sv. Sv. Kuzma and Damyan', OOD, Sofia
  - Medical Center Akademika EOOD, Sofia
  - Medical Center Hera EOOD, Sofia
  - Medical Center Intermedica, OOD, Sofia
  - Medical Center VAS OOD, Targovishte
  - DCC Mladost M - Varna, OOD, Varna
  - Mental Health Center-Vratsa EOOD, Vratsa
- India (19):
  - Local Institution - 616, Guwahati, Assam
  - Local Institution - 607, Ahmedabad, Gujarat
  - Local Institution - 604, Ahmedabad, Gujarat
  - Local Institution - 609, Surat, Gujarat
  - Local Institution - 613, Vadodara, Gujarat
  - Local Institution - 617, Belgavi, Karnataka
  - Local Institution - 614, Mangalore, Karnataka
  - Local Institution - 602, Mangalore, Karnataka
  - Local Institution - 601, Mysore, Karnataka
  - Local Institution - 611, Kozhikode, Kerala
  - Local Institution - 610, Aurangabad, Maharashtra
  - Local Institution - 619, Mumbai, Maharashtra
  - Local Institution - 603, Nagpur, Maharashtra
  - Local Institution - 608, Nashik, Maharashtra
  - Local Institution - 605, Nashik, Maharashtra
  - Local Institution - 615, Ajmer, Rajasthan
  - Local Institution - 618, Bikaner, Rajasthan
  - Local Institution - 606, Rajkot, Rajasthan
  - Local Institution - 612, Lucknow, Uttar Pradesh
- Japan (6):
  - Local Institution - 258, Kōnan, Aichi-ken
  - Local Institution - 250, Toyoake-shi, Aichi-ken
  - Local Institution - 257, Shirakawa, Fukushima
  - Local Institution - 254, Karatsu-shi, Saga-ken
  - Local Institution - 255, Fukuoka
  - Local Institution - 256, Tokyo
- Poland (9):
  - Local Institution - 506, Bialystok
  - Local Institution - 507, Gdansk
  - Local Institution - 509, Grudziądz
  - Local Institution - 501, Kielce
  - Local Institution - 503, Lodz
  - Local Institution - 505, Lublin
  - Local Institution - 502, Siemianowice Śląskie
  - Local Institution - 508, Suchy Las
  - Local Institution - 504, Tuszyn
- Romania (10):
  - Local Institution - 803, Brasov
  - Local Institution - 809, Bucharest
  - Local Institution - 804, Bucharest
  - Local Institution - 810, Bucharest
  - Local Institution - 802, Bucharest
  - Local Institution - 807, Bucharest
  - Local Institution - 808, Craiova
  - Local Institution - 801, Galati
  - Local Institution - 806, Iași
  - Local Institution - 805, Sibiu
- Serbia (12):
  - Clinical Center ' Dr Dragisa Misovic Dedinje', Belgrade
  - Institute of Mental Health, Belgrade
  - Local Institution - 413, Belgrade
  - Local Institution - 417, Belgrade
  - University Clinical Center of Serbia, Belgrade
  - "Special Hospital for Psychiatric Diseases ""Kovin""", Kovin
  - Special Hospital for Psychiatric Diseases 'Kovin', Kovin
  - University Clinical Center Kragujevac, Kragujevac
  - University Clinical Center Nis, Niš
  - Special Hospital for Psychiatric Diseases 'Gornja Toponica', Niš
  - Special Hospital for Psychiatric Diseases 'Sveti Vracevi', Novi Kneževac
  - Special Hospital for Psychiatric Disease 'Dr Slavoljub Bakalovic', Vršac
- United Kingdom (10):
  - Local Institution - 707, Pool, Reruth, Cornwall
  - Local Institution - 705, Brighton, East Sussex
  - Local Institution - 701, London, Greater London
  - Local Institution - 706, Ashton-under-Lyne, Greater Manchester
  - Local Institution - 710, Manchester, Greater Manchester
  - Local Institution - 709, Maidstone, Kent
  - Local Institution - 708, Oxford, Oxfordshire
  - Local Institution - 704, Glasgow, Strathclyde
  - Local Institution - 702, Chertsey, Surrey
  - Local Institution - 703, Birmingham, West Midlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com